CLINICAL TRIAL: NCT03291392
Title: CUHK Stroke Biobank
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Wai Hong Thomas, Professor, Chinese University of Hong Kong
Other Study IDs: crec no. 2014.582
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Ischemic; Genetic Disease; Atherosclerosis, Cerebral
Keywords: Genetics; Stroke; Biobank; Atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Genetic Diseases, Inborn; Intracranial Arteriosclerosis; Stroke; Atherosclerosis | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 30ml of EDTA blood, buccal swab or saliva, body tissue, or cerebrospinal fluid to be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atherosclerosis: Patient with intracranial stenosis or extracranial stenosis equal to or more than 70% would be invited to join the study for blood taking.
  Biobank: Gene expression or biomarkers exploration for atherosclerotic-related genetic diseases
  Interventions: Genetic: Gene expression or biomarkers exploration
- Family members: The stroke patient who had family history of stroke, their parents and siblings would also be invited to join the study for blood taking or buccal swab/ saliva collection.
  Biobank: Gene expression or biomarkers exploration for atherosclerotic-related genetic diseases
  Interventions: Genetic: Gene expression or biomarkers exploration
- Normal subjects: Normal subjects without ischemic stroke or intracranial/extracranial stenosis would be invited to join the study for blood taking.
  Biobank: Gene expression or biomarkers exploration for atherosclerotic-related genetic diseases
  Interventions: Genetic: Gene expression or biomarkers exploration

INTERVENTIONS:
Genetic: Gene expression or biomarkers exploration

SUMMARY:
The purpose of the study are:

1. To make quality, characterized samples and related data available for future studies, including Genome Wide Association Studies (GWAS), genomics, and biomarker research;
2. To use these samples and related medical information to answer research questions aimed at understanding the genetics and underlying biology of acquired disease and injury to the brain, heart and blood vessels with the express purpose of advancing the search for effective modalities for prevention, treatment, and recovery;
3. To develop additional operational infrastructure to support this project across the Prince of Wales Hospital and divisions, including (1) tracking of patient consent, (2) management of collection and sample processing processes, (3) sample inventory and QC/QA processes, and (4) release of materials to investigators for further research.

DETAILED DESCRIPTION:
TYPES OF TISSUES TO BE BANKED

Blood:

Blood will be collected from the out-patient clinic, prospectively at the time of a clinically planned procedure or prospectively during a procedure performed solely for research. After informed consent is obtained, the patient/ subject will be asked to donate a one-time blood sample of up to 30ml. A portion of each blood sample will be used to generate a DNA sample, and the remainder will be used to separate out plasma, peripheral blood cells, and/or serum for future research studies, including but not limited to metabolomics, proteomics, biomarker measurements, and bioenergetic assays.

Cerebrospinal Fluid:

Cerebrospinal fluid 5-10ml may be collected prospectively from lumbar puncture or the subset of patients who have an external ventricular drain (EVD) placed as part of their clinical care. The standard clinical protocol for EVD includes the drainage of CSF externally into a collection bag. Once the volume of CSF drainage is recorded, the CSF is typically discarded. The collection of CSF will be coordinated with the subject's primary treatment team. At this time, CSF banking will not occur in subjects who do not have CSF collection planned as part of their clinical care.

Body Tissue:

The body tissue will be collected from the patients who undergo the carotid stent which is their routine medical treatment. Around 5mg tissue will be taken from the filter wire during the stenting operation and then stabilized by RNAlater reagent immediately. The tissue will be kept in -80oC freezer for future process.

Buccal swab or saliva:

Buccal swab or saliva (~5-10ml) may be collected from the patients, their family members and/or normal subjects for DNA and RNA extraction if necessary. It would be collected by the trained doctor, medical staffs or research assistant. The collected samples will be kept in -80oC freezer for future use, for example, extraction of DNA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult equal or more 18 years of age and Chinese ONLY.
2. Stroke patients, their family members, and/or the normal subjects without intracranial stenosis or extracranial stenosis, are eligible to join the study.
3. Subject is willing to have blood taken, cerebral spinal fluid and/or body tissue drawn for storage in the research bank.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chinese ONLY
  2. Patients with intracranial stenosis or extracranial stenosis equal to or >70%
  3. Stroke patients and their family members
  4. Normal subject without any intracranial stenosis/ extracranial stenosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke-related genetics | Dec, 2025
  1. Discovery of novel genetic predictor of stroke and its complications will be done by identifying cases and controls for different stroke subtype and complications within the recruited samples, and using whole-genome genotyping arrays, or by sequencing approaches.
  2. Replication of novel genetic markers of stroke will be performed using a combination of genotyping, multiplex genotyping, customized-content genotyping arrays and sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wai Hong LEUNG, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Tissues and data from the repository will only be shared with other academic, non-profit institutions. No collaboration with for-profit companies is anticipated. All investigators seeking to gain access to the repository must first demonstrate that their research interests are relevant to the central theme of the repository. Investigators must also complete all required IRB documentation before samples and information will be released.
  In the event that a commercial, for-profit, collaboration is sought, a bona fide intellectual collaboration between the PI and an individual or group at the for-profit site and a Materials Transfer Agreement will be required. For all researchers requesting samples, the IRB recommended Letter of Agreement must be signed prior to our releasing tissues and information.